CLINICAL TRIAL: NCT01283464
Title: Double-blinded, Single-center, Parallel-arm Comparison Study of Retinol 1.0% and Tretinoin 0.02% in the Treatment of Moderate to Severe Photodamage
Brief Title: Comparison of Retinol 1.0% and Tretinoin 0.02% in the Treatment of Moderate to Severe Photodamage and Wrinkles
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Anna Chien, Assistant Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SKM10-R-01
Record Dates: First submitted 2011-01-24; First posted 2011-01-26 (Estimated); Results first posted 2013-08-20 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Photodamaged Skin; Wrinkles
Keywords: Retinol; Tretinoin
MeSH Terms: interventions — Vitamin A; Tretinoin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Retinol (Active Comparator): Retinol 1.0% cream
  Interventions: Drug: Retinol
- Tretinoin (Active Comparator): Tretinoin 0.02% cream
  Interventions: Drug: Tretinoin

INTERVENTIONS:
Drug: Retinol — 1.0% cream
  Arms: Retinol
Drug: Tretinoin — 0.02% cream
  Other Names: Retin-A; Renova; Atralin; Aberela; Airol; Avita; Stieva-A
  Arms: Tretinoin

SUMMARY:
The purpose of this study is to assess the comparative efficacy of retinol 1.0% and tretinoin 0.02% in minimizing wrinkles, discoloration, roughness, and other signs of moderate to severe photodamage. Our hypothesis is that both products will be of comparable benefit.

ELIGIBILITY:
Inclusion Criteria:

* Age 35 or over
* Moderate to severe photodamage

Exclusion Criteria:

* History of facial cosmetic surgery, facial resurfacing procedures, deep peels, or facial fillers
* History of keloids or hypertrophic scars
* Use of oral steroids or oral retinoids (such as Accutane) in past 6 months

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Dept. of Dermatology, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Chien AL, Kim DJ, Cheng N, Shin J, Leung SG, Nelson AM, Zang J, Suh H, Rainer B, Wallis L, Okoye GA, Loss M, Kang S. Biomarkers of Tretinoin Precursors and Tretinoin Efficacy in Patients With Moderate to Severe Facial Photodamage: A Randomized Clinical Trial. JAMA Dermatol. 2022 Aug 1;158(8):879-886. doi: 10.1001/jamadermatol.2022.1891. PMID 35675051
- See also: SkinMedica, Inc., company website — http://www.skinmedica.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study period: January 2011-December 2011 Recruitment period: January 2011-June 2011 Setting: Academic referral center
Groups:
- Retinol: Retinol 1.0% cream to entire face daily or as tolerated for 6 months
- Tretinoin: Tretinoin 0.02% cream to entire face daily or as tolerated for 6 months
Period: Overall Study
Arm/Group | Retinol | Tretinoin
Started | 12 | 12
Completed | 10 | 11
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Retinol | Tretinoin | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (11.3) | 62.7 (7.6) | 61.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Global Photodamage Severity
Description: A photonumeric scale for the assessment of cutaneous photodamage (CE Griffiths, et al). Five photographic standards (en face and 45 degrees oblique) illustrating increasing severity of photodamage (min=0, max=8) where 0=no damamge; 2=mild damage; 4=moderate damage; 6=moderate/severe damage; and grade 8=severe damage.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Retinol | Tretinoin
Number analyzed (Participants) | 12 | 12
units on a scale | 4.8 (1.687) | 5.45 (1.572)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Other (non-serious) Adverse Events were collected/assessed in the entire study population, but none observed. A total of 3 serious adverse events occurred during the course of the trial.
Arm/Group | Retinol | Tretinoin
Serious Adverse Events (participants affected / at risk) | 1/12 | 2/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retinol (N=12) | Tretinoin (N=12)
inpatient admission for pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
inpatient admission for orthopedic surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
inpatient admission for near syncopal episode (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No